CLINICAL TRIAL: NCT06074302
Title: Use of a Hyaluronic Acid Filler (Resilient Hyaluronic Acid [RHA] Redensity) for Improvement of Radial Cheek Lines
Brief Title: Hyaluronic Filler for Improvement of Radial Cheek Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Main Line Center for Laser Surgery (Other)
Responsible Party: Principal Investigator, Kachiu Lee, MD, Physician, Main Line Center for Laser Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHA10823
Record Dates: First submitted 2023-07-27; First posted 2023-10-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment of radial cheek lines with RHA Redensity (Experimental): A total of 20 patients with facial fine lines of the cheeks/radial cheek lines will be treated with RHA Redensity. They will receive 2 treatments.
  During the first treatment visit, up to 2cc of RHA Redensity will be injected in a microdroplet technique per cheek. The boundaries of the injection area will be defined by the nasolabial fold, nasojugal groove, palpebromalar groove, mandible, and preauricular crease. Patients will return in 4 weeks for another treatment visit using the same technique. At 8 weeks, they will return for a follow-up visit.
  Interventions: Device: RHA Redensity

INTERVENTIONS:
Device: RHA Redensity — RHA Redensity will be injected in a microdroplet technique to bilateral cheeks.

SUMMARY:
Appearance of superficial radial cheek lines and fine lines of the cheek are signs of photoaging. These lines appear in a curvilinear or crosshatched fashion on the lower cheeks in photoaged individuals. They represent a common concern among patients seeking cosmetic treatments. With the aging population and increasing social awareness of cosmetic treatments, it is likely that the demand for filler procedures will increase. Current treatment options for these lines include fractionated and fully ablative laser resurfacing, topical retinoids, intradermal filler injections, and chemical peels.

One potential treatment for facial fine lines include use of low G' hyaluronic acid fillers, which allow for dynamic movement while also addressing the appearance of the lines. Resilient Hyaluronic Acid (RHA) Redensity is an FDA-cleared filler used for treatment of dynamic perioral rhytids. Hyaluronic acid-based fillers have been shown to improve overall skin texture (skin surface hydration, roughness, and elasticity) through the hypothesized mechanism of inducing a fibroblast response to boost collagen production. They have the potential to reduce appearance of facial fine lines of the cheek. This study will evaluate the efficacy of RHA Redensity in improving radial cheek lines.

DETAILED DESCRIPTION:
This clinical investigation is a prospective study consisting of a 2 treatment visits and a follow-up visit. A total of 20 patients will be recruited.

Treatment Plan Screening Visit and Treatment Visit 1 A total of 20 patients with facial fine lines of the cheeks/radial cheek lines will be treated with Resilient Hyaluronic Acid (RHA) Redensity, off-label. Patients will be consented, photographed with the Canfield Visia, and be asked to fill out the Facial Appearance, Health-Related Quality of Life and Adverse Effects (FACE-Q) Appraisal of Lines: Overall and FACE-Q Age Appraisal Visual Analog Scale surveys. The physician will fill out the Allergan Fine Lines Scale.

After discussion with the patient, volume of filler needed will be determined at the discretion of the provider, up to 2cc per cheek. RHA Redensity will be applied using a microdroplet technique, with approximately 0.02-0.04cc of product injected sub-dermally approximately 0.5-1cm apart on the malar and nasolabial cheek. The boundaries of the injection area will be defined by the nasolabial fold, nasojugal groove, palpebromalar groove, mandible, and preauricular crease. After treatment, the area will be lightly massaged by the physician. The patient will be asked to ice the area 3 times daily for 24 hours and post-op instructions will be provided.

Treatment Visit 2 (4 weeks +/- 2 weeks) Photographs using the Canfield Visia will be taken. Patients will return for a repeat treatment of RHA Redensity of the cheek using the microdroplet technique as described above. A maximum of 2cc will be used per cheek.

Follow-up visit (8 weeks +/-2 weeks) Patients will be photographed and will be asked to fill out the FACE-Q Appraisal of Lines: Overall and FACE-Q Age Appraisal Visual Analog Scale surveys. The physician will fill out the Allergan Fine Lines Scale. The patient will fill out the FACE-Q Appraisal of Lines: Overall and FACE-Q Age Appraisal Visual Analog Scale surveys. Photographs of the patient will be captured using the Canfield Visia camera.

ELIGIBILITY:
Inclusion Criteria:

* 31 years old or great
* Rating of 2, 3, or 4 on 5-point Allergan Fine Lines Scale on the cheeks

Exclusion Criteria:

* Pregnancy
* Prior adverse reaction to hyaluronic acid treatment (injectable or over-the-counter topical)
* Connective tissue disorder
* Active infection in treatment area
* Active severe inflammatory disease in treatment area such as atopic dermatitis, psoriasis
* Treatment with toxin or filler in lower face below the orbital rim within the past 6 months

Min Age: 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Allergan Fine Lines Scale | 10 weeks
  1-point improvement of facial fine lines of the cheek based on the validated Allergan Fine Lines Scale between baseline and 8-week follow-up. Scale is a 5-point scale rated from 0 to 4, with 0 representing no fine lines and 4 representing diffuse fine lines with cross-hatching.

SECONDARY OUTCOMES:
FACE-Q Appraisal of Lines: Overall | 10 weeks
  Improvement in scores in patient-reported outcomes based on the validated FACE-Q Appraisal of Lines: Overall between baseline and 8-week follow-up. Scale is scored on a 1-100 scale, with 100 representing excellent quality of life with regards to facial fine lines.

CONTACTS AND LOCATIONS:
Overall Officials: Kachiu Lee, Principal Investigator — Physician
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alzahrani F, Alajmi A, Lee KC. A Dynamic, High-Stretch Resilient Hyaluronic Acid Filler Improves Fine Lines of the Cheek and Patient-Reported Outcomes. Dermatol Surg. 2025 Mar 26;51(8):773-777. doi: 10.1097/DSS.0000000000004625. PMID 40135789